CLINICAL TRIAL: NCT01090726
Title: Intubation With Storz Videolaryngoscope® Versus Airtraq® - in an Infant Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Martin Kryspin Soerensen/ MD, Department of Anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1A-INF-STORZ-AIR
Record Dates: First submitted 2010-03-18; First posted 2010-03-22 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-03

CONDITIONS: Intubation; Videolaryngoscopy; Infant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Storz videolaryngoscope (Experimental): Macintosh overview followed by Airtraq overview followed by Storz videolaryngoscope overview and intubation.
  Interventions: Device: Storz videolaryngoscope
- Airtraq (Active Comparator): Macintosh overview followed by Storz videolaryngoscope overview followed by Airtraq overview and intubation.
  Interventions: Device: Airtraq

INTERVENTIONS:
Device: Storz videolaryngoscope — Storz videolaryngoscope being used for the actual intubation
  Arms: Storz videolaryngoscope
Device: Airtraq — Airtraq being used for the actual intubation
  Arms: Airtraq

SUMMARY:
The purpose of the pilot study is to compare new laryngoscopes for infants by assessing the equipment best suited to assist the intubation, with the best overview, shortest time to intubation and use these numbers to make a sample size calculation for the full protocol. The investigators hypothesis is that the Storz videolaryngoscope® has a better success rate than infants (<2 years). The patients will be optimally anaesthetized with neuromuscular blockade for the intubation. All patient will be evaluated with af Macintosh blade laryngoscope, with an Airtraq® or a Storz videolaryngoscope®, and finally intubated with the other one of the later, which the patient was randomized to.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical patients ASA-class 1-2 below the age of 2 years, with indication for intubation.
* Informed consent from parent.
* The parents must have legal custody of the child.
* The parents must be able to read and understand Danish.

Exclusion Criteria:

* Expected difficult airway.

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Success rate | 5 minutes
  Succes is defined by intubation being executed in the first try.

SECONDARY OUTCOMES:
Time to Cormack evaluation | 5 minutes
Time to intubation | 5 minutes
Number of intubation attempts | 5 Minutes
Quality of laryngeal overview before intubation | 5 Minutes
  Evaluated by Cormack score
Prevalence of post intubation stridor | 12 hours
Intubation conditions | 5 Minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesia, Centre of Head and Orthopaedics, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Lingappan K, Neveln N, Arnold JL, Fernandes CJ, Pammi M. Videolaryngoscopy versus direct laryngoscopy for tracheal intubation in neonates. Cochrane Database Syst Rev. 2023 May 12;5(5):CD009975. doi: 10.1002/14651858.CD009975.pub4. PMID 37171122
- [Derived] Sorensen MK, Holm-Knudsen R. Endotracheal intubation with airtraq(R) versus storz(R) videolaryngoscope in children younger than two years - a randomized pilot-study. BMC Anesthesiol. 2012 Apr 30;12:7. doi: 10.1186/1471-2253-12-7. PMID 22545575